CLINICAL TRIAL: NCT07340008
Title: Comparison of Intramuscular Ketamine and Intranasal Nalbuphine and Dexmedetomidine for Analgosedation in Children Undergoing Suture Removal After Surgery for Congenital Clefts of the Palate, Alveolar Ridge, and Lip
Brief Title: Analgosedation With Ketamine, Nalbuphine, or Dexmedetomidine for Suture Removal in Children After Cleft Surgery
Acronym: KID-CLEFT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKCLJ-KID-CLEFT-TP 20240163; TP 20240163 (Other Grant/Funding Number: University Medical Centre Ljubljana - Tertiary Research Fund)
Record Dates: First submitted 2025-08-27; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-10

CONDITIONS: Orofacial Clefts; Cleft Lip and Palate; Alveolar Ridge Defect
Keywords: pediatric sedation; Cleft surgery; Ketamine; Dexmedetomidine; Nalbuphine; Intranasal sedation; Intramuscular injection; Sedation in children
MeSH Terms: conditions — Cleft Lip | interventions — Ketamine; Nalbuphine; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Parallel assignment with three intervention arms. Children aged 6 months to 3 years undergoing suture removal after cleft surgery will be randomly assigned to receive one of the following for procedural sedation: intramuscular ketamine, intranasal nalbuphine, or intranasal dexmedetomidine. The study will compare onset, depth, and duration of sedation, surgeon-rated ease of procedure, recovery time, and safety profiles of each drug.
Masking Description: This is an open-label study. No participants, investigators, or outcome assessors are blinded to the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intramuscular Ketamine (Active Comparator): Participants assigned to this arm will receive intramuscular ketamine at a dose of 4 mg/kg body weight for analgosedation during suture removal after surgery for congenital clefts. In addition, glycopyrrolate 4 mcg/kg will be administered intramuscularly to reduce salivation. This arm represents the control group, following the established clinical protocol.
  Interventions: Drug: ketamine
- Intranasal Nalbuphine (Experimental): Participants assigned to this arm will receive intranasal nalbuphine at a dose of 0.5 mg/kg body weight, administered using a mucosal atomizer device (MAD), for analgosedation during suture removal after cleft surgery. This intervention will be evaluated for its effectiveness, ease of administration, and safety compared with intramuscular ketamine.
  Interventions: Drug: Nalbuphine
- Intranasal Dexmedetomidine (Experimental): Participants assigned to this arm will receive intranasal dexmedetomidine at a dose of 3 mcg/kg body weight, administered using a mucosal atomizer device (MAD), for analgosedation during suture removal after cleft surgery. The intervention will be evaluated for sedation depth, response to separation from parents, and overall procedural ease compared with other sedative agents.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: ketamine — Intramuscular administration of Ketamine at 4 mg/kg body weight for analgosedation during suture removal in children after surgery for congenital clefts. Glycopyrrolate 4 mcg/kg will be co-administered to reduce salivation.
  Other Names: Ketamine Hydrochloride; Ketanest; Ketalar
  Arms: Intramuscular Ketamine
Drug: Nalbuphine — Intranasal administration of Nalbuphine at 0.5 mg/kg body weight via mucosal atomizer device (MAD) for analgosedation during suture removal after cleft surgery in children.
  Other Names: Nalbuphine Hydrochloride; Nubain
  Arms: Intranasal Nalbuphine
Drug: Dexmedetomidine — Intranasal administration of Dexmedetomidine at 3 mcg/kg body weight via mucosal atomizer device (MAD) for analgosedation during suture removal after cleft surgery in children.
  Other Names: Dexmedetomidine Hydrochloride; Precedex; Dexdor
  Arms: Intranasal Dexmedetomidine

SUMMARY:
This prospective, randomized study is designed to compare the efficacy and safety of three sedative-analgesic agents-intramuscular ketamine, intranasal nalbuphine, and intranasal dexmedetomidine-for procedural sedation in children undergoing suture removal following cleft palate, alveolar ridge, or lip surgery. The study will include 60 children aged 6 months to 3 years, randomly assigned to one of three intervention groups.

The primary objectives are to compare time to achieve adequate sedation (Modified Ramsay Sedation Scale 2-3), surgeon-rated ease of surgical procedure, and time to discharge readiness (Modified Aldrete Score ≥9). Secondary outcomes include baseline child behavior, response to drug administration, depth of sedation, response to separation from parents, and parental satisfaction, as well as monitoring of perioperative complications and vital signs.

All study medications are approved and commonly used in pediatric anesthesia. The trial will be conducted using non-invasive monitoring, with intravenous access established only in case of emergency interventions. Findings from this study are expected to provide evidence to optimize pediatric sedation protocols for minor surgical procedures.

DETAILED DESCRIPTION:
Title: Comparison of Intramuscular Ketamine and Intranasal Nalbuphine and Dexmedetomidine for Analgosedation in Children Undergoing Suture Removal After Surgery for Congenital Clefts of the Palate, Alveolar Ridge, and Lip

Introduction Orofacial clefts, including cleft lip with or without cleft palate and isolated cleft palate, are among the most common congenital craniofacial anomalies. Primary correction of a cleft lip may be performed between the 6th week and the 6th month of life, considering the child's growth, identification of associated anomalies, and avoidance of general anesthesia in the neonatal period. In cases of congenital cleft palate or alveolar ridge, correction is typically completed between 6 and 12 months of age.

Suture removal following these surgeries is a short procedure that requires optimal sedation and analgesia to enable efficient, rapid, and safe completion. The American College of Emergency Physicians (ACEP) defines procedural sedation as "a technique of administering sedatives or dissociative agents with or without analgesics to facilitate a procedure while maintaining cardiorespiratory function." The goal of sedation in pediatric patients is to avoid fear of medical professionals, injections, surgery, and the operating room environment. Effective sedation improves safety and comfort, reduces pain and anxiety, enhances the possibility of amnesia, and minimizes psychological trauma from separation from parents and exposure to an unfamiliar environment.

Ketamine is a dissociative anesthetic and analgesic, an NMDA receptor antagonist synthesized in 1962. It is favored for its analgesic and amnestic effects, preservation of airway reflexes, and various routes of administration (IV, IM, oral, rectal, nasal, epidural, intrathecal). However, ketamine may cause unpleasant hallucinations and hypersalivation. It is relatively contraindicated in patients with hypertension, increased intracranial pressure, respiratory infections, or underlying neuropsychiatric disorders.

Dexmedetomidine, approved by the FDA in 1999, is a selective α2-adrenoceptor agonist with strong sedative, analgesic, and anxiolytic properties, commonly used in pediatric intensive care units and diagnostic/therapeutic procedures. It may cause hypotension and bradycardia. Literature describes its pediatric use in intraoperative sedation, delirium management, postoperative analgesia, and shivering prevention.

Nalbuphine hydrochloride is a kappa-opioid receptor agonist and partial mu-antagonist. It exhibits a "ceiling effect," preventing respiratory depression. Nalbuphine is safe and effective for pediatric analgesia and sedation, and is administered via subcutaneous, IM, IV, or intranasal routes. Atomized intranasal delivery, using a Mucosal Atomizer Device (MAD), avoids painful IV access, offering a simple, safe, and effective method.

This study is designed to compare three sedatives-ketamine, dexmedetomidine, and nalbuphine-in children undergoing suture removal after cleft surgeries, focusing on perioperative sedation quality, procedural ease, application convenience, and safety profiles.

Protocol This prospective, randomized study will be conducted at the Department of Maxillofacial and Oral Surgery, University Medical Centre Ljubljana, in collaboration with anesthesiologists and surgeons.

A total of 60 children aged 6 months to 3 years requiring suture removal after cleft surgeries will be enrolled. Exclusion criteria include known allergy to the study drugs, ASA status greater than II, and lack of informed parental consent. After completion of the consent process, patients will be randomized into three groups.

Premedication with midazolam will be administered 30 minutes before the procedure. Group 1 will receive intramuscular ketamine (4 mg/kg) plus glycopyrrolate (4 mcg/kg) to reduce salivation. Group 2 will receive intranasal nalbuphine (0.5 mg/kg), and Group 3 intranasal dexmedetomidine (3 mcg/kg), delivered via MAD. Due to the short duration of the procedure and minimal risk, IV access will not be established unless complications arise.

If sedation is insufficient to complete the procedure, inhaled sevoflurane (starting at 2%, titrated by 0.5% increments) will be used as rescue medication.

Vital signs (heart rate, oxygen saturation, non-invasive blood pressure) will be monitored continuously. Blood pressure will be recorded three times: before drug administration, during the procedure, and prior to discharge. Additional monitoring will occur in case of adverse events. Heart rate and oxygen saturation will be recorded every 5 minutes before surgery, every 2 minutes during the procedure, and every 5 minutes post-procedure until discharge.

Sedation onset time, procedure duration, and recovery time will be evaluated. Complications (e.g., bronchospasm, aspiration, laryngospasm) will be documented, along with sedation depth (Modified Ramsay Scale), child's response to separation from parents, and surgeon-rated ease of procedure.

Statistical Methods It is expected that ketamine will demonstrate the fastest onset, dexmedetomidine the longest duration and calmest effect, and nalbuphine the most stable hemodynamics. Statistical analysis will include the Shapiro-Wilk test for normality. Normally distributed data will be expressed as mean ± SD, and non-normal data as median (IQR). Categorical variables will be presented as frequencies (%). Kruskal-Wallis test, Fisher's exact test, and Dunn's post-hoc test will be applied as appropriate. A p-value < 0.05 will be considered statistically significant. Analyses will be performed using SPSS 13.0 (SPSS Inc., Chicago, IL, USA).

ELIGIBILITY:
Inclusion criteria:

* Age 6 months to 3 years
* Scheduled for suture removal after surgery for congenital cleft of the palate, alveolar ridge, or lip
* American Society of Anesthesiologists (ASA) physical status I or II
* Written informed consent obtained from parents or legal guardians
* Slovene-speaking family to ensure understanding and compliance
* No contraindications to the use of study medications

Exclusion criteria:

* Known allergy or hypersensitivity to ketamine, nalbuphine, or dexmedetomidine
* ASA physical status greater than II
* Significant neurological, psychiatric, or respiratory disorder
* Active or recent upper respiratory tract infection
* Refusal of parental or guardian consent
* Developmental disorder affecting communication or cooperation

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Time to achieve adequate sedation (Modified Ramsay Sedation Score 2-3) | Perioperatively, from drug administration until Modified Ramsay score 2-3 is achieved (typically within 5-20 minutes)
  Time in minutes from administration of the study drug until the child reaches adequate sedation, defined as a Ramsay Sedation Score of 2-3. Sedation is assessed every 5 minutes by a trained clinician.
  Unit of Measure: Minutes
Sedation depth before procedure (Modified Ramsay Sedation Scale) | Periprocedural (every 5 minutes for up to 20 minutes after study drug administration, until procedure begins)
  Sedation depth is measured using the Modified Ramsay Sedation Scale (1 = anxious/agitated, 6 = no response; 2-3 = adequate sedation). A trained clinician assesses sedation every 5 minutes after administration of the study drug, until the start of the suture removal procedure.
Surgeon-rated ease of surgical procedure | Within 5 minutes after completion of suture removal
  Ease of suture removal as rated by the operating surgeon using a 5-point Likert scale (1 = very difficult, 5 = very easy).
  Unit of measure: Units on a scale
Time to discharge from recovery room | Perioperative (every 5 minutes post-procedure until Modified Aldrete Score ≥9 is achieved or until discharge from the recovery area, up to 90 minutes)
  Time in minutes from the end of the surgical procedure until the child reaches a Modified Aldrete Score of ≥9, indicating readiness for discharge from the recovery area to the hospital ward. The Aldrete score is assessed every 5 minutes by recovery room nursing staff.
  Unit of Measure: Minutes
Discharge readiness (Modified Aldrete Score) | Postprocedural (every 5 minutes in recovery room until Modified Aldrete Score ≥9 is reached, up to 90 minutes post-procedure)
  Discharge readiness assessed using the Modified Aldrete Score (range: 0-10; score ≥9 indicates clinical criteria for transfer to ward).
  Unit of Measure: Units on a scale

SECONDARY OUTCOMES:
Baseline child behavior (Ohio Behavioral Rating Scale) | Baseline (within 5 minutes prior to study drug administration during the procedure)
  Child's baseline behavior assessed using the Ohio Behavioral Rating Scale (1 = calm/cooperative, 4 = combative/uncontrollable; higher scores = more difficult behavior).
  Unit of measure: Units on a scale
Child's response to drug administration | Periprocedural (immediately during study drug administration)
  Child's behavioral response during study drug administration, assessed using a 4-point scale (1 = calm acceptance, 4 = severe resistance; higher scores = greater resistance).
  Unit of measure: Units on a scale
Child's behavior during separation from parent | Periprocedural (immediately at the time of parent-child separation)
  Behavior assessed on a 4-point separation scale (1 = excellent/easy separation, 4 = poor/difficult separation; higher scores indicate greater distress).
  Unit of measure: Units on a scale
Use of rescue Sevoflurane due to inadequate sedation | Intraoperatively, during the suture removal procedure
  Number of participants who required additional sedation using inhaled Sevoflurane due to inadequate procedural sedation or significant patient movement during suture removal.
  The rescue protocol includes Sevoflurane inhalation starting at 2% concentration via facemask, with titration increased by 0.5% every minute as needed, until adequate sedation is achieved to complete the procedure safely.
  The indication for administration is failure to maintain adequate sedation (Modified Ramsay Sedation Scale <2 or excessive movement interfering with surgery), as assessed by the attending anesthesiologist.
  Unit of Measure: Number of participants
Sedation level measured by Modified Ramsay Sedation Scale during procedure | From drug administration until end of suture removal procedure (expected duration up to 30 minutes)
  Sedation level will be assessed using the Modified Ramsay Sedation Scale (range: 1-6; higher scores indicate deeper sedation). The target for adequate sedation is defined as a score of 2-3.
  Sedation scores will be recorded:
  * every 5 minutes from study drug administration until start of procedure,
  * and then every 2 minutes during the procedure until completion of suture removal.
  This outcome complements the primary endpoint "Time to achieve adequate sedation (Ramsay 2-3)" by describing the actual sedation scores across time points.
  Unit of Measure: Units on a scale
Parental satisfaction with sedation | Collected immediately after completion of procedure.
  Parental satisfaction with the sedation process, assessed using a 5-point Likert scale (1 = very dissatisfied, 5 = very satisfied).
  Unit of measure: Units on a scale

OTHER OUTCOMES:
Heart rate monitoring | From study drug administration until discharge from recovery room (up to 90 minutes)
  Heart rate (HR) will be continuously monitored and recorded every 5 minutes during sedation, every 2 minutes during the procedure, and every 5 minutes in the recovery area.
  Unit of Measure: Beats per minute (bpm)
Blood pressure monitoring | From baseline (pre-sedation) to discharge readiness (within 90 minutes post-procedure)
  Systolic and diastolic blood pressure will be measured at three key time points: before sedation, during the procedure, and prior to discharge. Additional measurements will be taken in case of complications.
  Unit of Measure: mmHg
Oxygen saturation monitoring | From study drug administration until discharge from recovery room (up to 90 minutes).
  Oxygen saturation (SpO₂) will be monitored continuously using pulse oximetry and documented every 5 minutes during sedation and recovery, and every 2 minutes during the procedure.
  From study drug administration until disch Unit of Measure: Percentage (%)
Respiratory rate monitoring | From baseline until discharge from recovery room (up to 90 minutes)
  Respiratory rate will be observed and recorded at baseline, during the procedure, and in the recovery area every 5 minutes.
  Unit of Measure: Breaths per minute
Incidence of laryngospasm | Periprocedural period (from study drug administration to discharge from the recovery room)
  Number of participants who experience laryngospasm during the perioperative period, assessed clinically by anesthesiology staff.
  Unit of Measure: Number of participants
Incidence of bronchospasm | Periprocedural period (from study drug administration to discharge from the recovery room)
  Number of participants who experience bronchospasm, confirmed by auscultation and clinical observation.
  Unit of Measure: Number of participants
Incidence of apnea | During procedure and recovery phase (up to 90 minutes after drug administration).
  Description:
  Number of participants with observed episodes of apnea (>20 seconds pause in breathing).
  Unit of Measure: Number of participants
Incidence of desaturation | Periprocedural period (from study drug administration to discharge from recovery room)
  Number of participants with oxygen saturation <90% at any point during the procedure or recovery, measured via pulse oximetry.
  Unit of Measure: Number of participants
Incidence of postoperative nausea and vomiting (PONV) | Perioperative/Periprocedural (i.e., from the administration of the study drug until discharge from the recovery area, covering the entire period during which postoperative nausea and vomiting may occur)
  Number of participants with reported or observed nausea or vomiting during recovery.
  Unit of Measure: Number of participants
Incidence of agitation | Perioperative/Periprocedural (i.e., from the end of the procedure until discharge from the recovery area, capturing the full recovery phase during which agitation may occur)
  Number of participants showing signs of emergence agitation, defined by physical restlessness or inconsolable crying during recovery.
  Unit of Measure: Number of participants
Total number of perioperative complications per treatment group | Perioperative/Periprocedural (i.e., from study drug administration until discharge from the recovery room)
  Total number of recorded perioperative complications in each treatment group (Ketamine, Nalbuphine, Dexmedetomidine), regardless of type or severity. One participant may contribute multiple events.
  Unit of Measure: Number of complications
Mean number of complications per participant | Perioperative/Periprocedural (i.e., from study drug administration until discharge from the recovery room)
  Average number of complications experienced per participant in each group, calculated by dividing total complications by number of participants in that group.
  Unit of Measure: Number of complications per participant
Severity grading of perioperative complications | Perioperative/Periprocedural (i.e., from study drug administration until discharge from the recovery room)
  Severity of each complication will be assessed and classified as mild, moderate, or severe according to predefined clinical criteria. The distribution of severity grades will be analyzed across treatment groups.
  Number of events by severity level (mild/moderate/severe).

CONTACTS AND LOCATIONS:
Overall Officials: Tadej P Dovšak, DDS, MD, PhD, Study Chair — University Medical Centre Ljubljana, Department of Maxillofacial and Oral Surgery
Locations (1):
- Department of Maxillofacial and Oral Surgery, University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The dataset includes sensitive health information of pediatric participants. Due to ethical considerations and data protection regulations, data sharing is not planned within the scope of this study.